CLINICAL TRIAL: NCT01013103
Title: Effects of Atorvastatin on Endothelial Function, Vascular and Myocardial Redox State in High Cardiovascular Risk Patients
Brief Title: Pleiotropic Effects of Atorvastatin in High Cardiovascular Risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Dimitris Tousoulis, Professor of Cardiology, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AT-1002009
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease; HMG-CoA Reductase Inhibitor Toxicity; Atherosclerosis; Oxidative Stress; Endothelial Dysfunction
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin, Ischemic Heart Disease (Other)
  Interventions: Drug: Atorvastatin, high vs low dose
- Atorvastatin vs Placebo Cardiac Surgery (Placebo Comparator)
  Interventions: Drug: Atorvastatin vs Placebo

INTERVENTIONS:
Drug: Atorvastatin, high vs low dose — In this arm patients with ischemic heart disease will be recruited. In a double-blind crossover design heart failure patients (n=30) naïve to statins treatment will be randomized to receive oral atorvastatin 10mg/day 1x1(n=15) or oral atorvastatin 40mg/day 1x1 (n=15) for 4 weeks. At the end of 4 weeks a 2-week wash out period will follow and then all patients will switch atorvastatin dose and continue treatment for 4 weeks (e.g all patients that were under atorvastatin 10mg/day will be switched to atorvastatin 40mg/day and vice versa).
  Other Names: Atorvastatin high vs low dose in ischemic heart disease
  Arms: Atorvastatin, Ischemic Heart Disease
Drug: Atorvastatin vs Placebo — In this arm, patients undergoing cardiac surgery (CABG, valve replacement or aortic surgery) that are not under statins treatment will be recruited. Patients will be randomized in a double-blind fashion to atorvastatin 40mg/day or placebo for 3 days before surgery date.
  Other Names: Atorvastatin in Patients Undergoing Cardiac Surgery
  Arms: Atorvastatin vs Placebo Cardiac Surgery

SUMMARY:
The present study constitutes a study examining the effect of atorvastatin on vascular function in high cardiovascular risk patients. For this purpose the investigators will record atorvastatin effects on statin-naïve patients (patients that start statins treatment for first time). More specifically the investigators will study atorvastatin effects on:

1. Endothelial function
2. Arterial elastic properties
3. Systemic Inflammatory/thrombotic mechanisms
4. Vascular and myocardial redox state

DETAILED DESCRIPTION:
In total we will recruit 72 high cardiovascular risk patients such as patients with ischemic cardiomyopathy (ischemic heart failure), coronary artery disease and/or patients undergoing elective coronary bypass artery grafting (CABG), valve replacement or aortic surgery. The whole study will be divided into 2 distinct clinical arms:

ARM A

In this arm patients with ischemic heart failure (NYHA II-III) will be recruited. In a double-blind crossover design heart failure patients (n=30) naïve to statins treatment will be randomized to atorvastatin 10mg/day (n=15) or 40mg/day (n=15) for 4 weeks. At the end of 4 weeks a 2-week wash out period will follow and then all patients will switch atorvastatin dose (e.g all patients that were under atorvastatin 10mg/day will be switched to 40mg/day and vice versa).

Both at baseline and at the end of 4 weeks period patients will undergo

* blood sampling
* assessment of endothelium-dependent and -independent vasodilatation and
* vascular elastic properties study (see below for methods).

ARM B

In this arm, patients undergoing cardiac surgery (CABG, valve replacement or aortic surgery) that are not under statins treatment will be recruited (n=42). Patients will be randomized in a double-blind fashion to atorvastatin 40mg/day or placebo for 3 days before surgery.

Both at baseline and on surgery day patients will undergo

* blood sampling and
* assessment of endothelium-dependent and -independent vasodilatation (see below for methods) while
* during surgery tissue samples (grafts, myocardium and adipose tissue segments) will be obtained that will be used for ex-vivo studies (see below).

Consent form

Every patient participating in the clinical study will give a written consent form, and will be informed in details for the aims of the study by the researchers. During recruitment process all participants will fill out a questionnaire with demographic and clinical data. All information given by the participants will be held highly classified. All participants will give written consent for the programmed biochemical measurements and vascular studies, as stated in the study design. Specifically for patients undergoing cardiac surgery (arm B) an additional consent form will be filled out that will permit grafts, myocardium and adipose tissue segments harvesting during cardiac surgery.

Methods

Endothelial-dependent and independent vasodilatation: Brachial Artery Flow-Mediated Dilatation (FMD) of the brachial artery will be measured as a quantitative readout of NO-mediated conduit vessel endothelial function, as we have done in several previous studies and in accordance with international guidelines.Endothelial dependent (hyperaemic flow after cuff occlusion) and endothelial independent (GTN) responses of the brachial artery will be measured using high-resolution ultrasound imaging with automated vessel diameter measurements (Vascular Analyser, MIA Inc. Iowa). FMD and GTN induced dilatation will be measured as absolute and proportional changes in arterial diameter.Reproducibility data from our laboratory show a coefficient of variation for inter-study measurements of <10% comparable to other reports.

Arterial Stiffness: Measures of central arterial stiffness are independent predictors of cardiovascular outcomes in large prospective studies and is inversely correlated with measures of endothelial function.Arterial tonometry is a simple, reproducible method to measure, non-invasively, arterial stiffness. We have already established measures of central aortic stiffness - augmentation index and aortic pulse wave velocity - using the Sphygmocor system for applanation tonometry (AtCor Medical, Australia). Mathematical transformation of the radial pulse waveform is used to derive the augmentation index.The difference in time for the pulse waveform to reach the carotid compared to the femoral artery measures pulse wave velocity down the aorta, with faster transit associated with a 'stiffer' aorta.

Systemic oxidative stress: We will study statins effects on systemic oxidative stress using a systemic oxidative stress marker like lipid peroxides. In more details lipid peroxides will be quantified in patients' plasma using malondialdehyde assay (ΜDA-TBARS).

Vascular oxidative stress: ROS generation in the vascular segments obtained during CABG will be determined by lucigenin-enhanced chemiluminescence. The same measurements will also be performed in myocardium segments obtained during CABG form the site of right atrium incision, where extracorporeal circulation cannula is inserted. Our aim is to determine statins effects on vascular and myocardial ROS generation.

Adipose tissue cultures: During cardiac surgery adipose tissue samples will be collected. In more details subcutaneous adipose tissue will be collected from the site of sternum incision; pericardial adipose tissue will be collected from the site close to right ventricle; and femoral adipose tissue will be collected from the area of saphenous vein harvesting (when available). Adipose tissue samples obtained during surgery will be cultured ex-vivo using a standard adipose tissue protocol.

Biochemical and inflammatory markers: Apart from the common laboratory screening tests (whole blood count, AST, ALT, γGT, ALP, Urea, Creatinine, glucose, total cholesterol, triglycerides, LDL, HDL, Na+, K+, Ca2+, CRP), we will determine additional proinflammatory and prothrombotic biomarkers in patients' plasma. More specifically, using enzyme-linked immunosorbent assay (ELISA) we will quantify interleukin-6 and other adipokines both in patients plasma and adipose tissue cultures supernatants. Using high precision liquid chromatography (HPLC) we will quantify biopterin plasma and vascular levels (tetrahydrobiopterin, dihydrobiopterin and total biopterins).Studies have shown that the abovementioned markers may have a prognostic value in high cardiovascular risk patients.

Statistical Analysis: Statistical analysis of results will be done separately according to the clinical group studied. Therefore there will be separate statistical analysis for ischemic heart failure patients group (arm A) and for the patients undergoing cardiac surgery (arm B). Especially for arm B we will compare reactive oxygen species generation from vascular wall and myocardium between patients randomized to placebo or atorvastatin 40mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease confirmed by coronary angiography.
* Patients undergoing cardiac surgery such as elective coronary bypass artery grafting (CABG), valve replacement or aortic surgery.
* All patients will not be under statins treatment for at least 6 months before their inclusion to the study.

Exclusion Criteria:

* Acute coronary syndrome during the last 2 months
* Renal failure (creatinine > 2,2 mg/dl)
* Severe liver disease. Prospective follow-up of liver enzymes will be performed by the physicians in charge, as indicated by the relative guidelines regarding statins use and according to the current clinical practice.
* Any chronic/acute inflammatory disease, autoimmune disease and/or cancer
* Use of anti-inflammatory drugs or vitamins supplements

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Vascular Nitric oxide bioavailability (Arm A + B) | At the start and at the end of 2-week treatment period (arm A) and at the start and at the end of 3-day treatment period (arm B)

SECONDARY OUTCOMES:
Vascular Redox state (Arm B) | At the end of 3-day treatment period
Myocardial redox state (Arm B) | At the end of 3-day treatment period
Systemic inflammatory, thrombotic and oxidative stress status (Arms A + B) | At the start and at the end of 2-week treatment period (arm A) and at the start and at the end of 3-day treatment period (arm B)
Vascular elastic properties (Arm A) | At the start and at the end of 2-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Tousoulis, Principal Investigator — Professor, Athens University Medical School
Locations (1):
- Hippocration Hospital, Athens University Medical School, Athens, Attica, Greece

REFERENCES:
- [Derived] Antoniades C, Demosthenous M, Reilly S, Margaritis M, Zhang MH, Antonopoulos A, Marinou K, Nahar K, Jayaram R, Tousoulis D, Bakogiannis C, Sayeed R, Triantafyllou C, Koumallos N, Psarros C, Miliou A, Stefanadis C, Channon KM, Casadei B. Myocardial redox state predicts in-hospital clinical outcome after cardiac surgery effects of short-term pre-operative statin treatment. J Am Coll Cardiol. 2012 Jan 3;59(1):60-70. doi: 10.1016/j.jacc.2011.08.062. PMID 22192670
- [Derived] Antoniades C, Bakogiannis C, Leeson P, Guzik TJ, Zhang MH, Tousoulis D, Antonopoulos AS, Demosthenous M, Marinou K, Hale A, Paschalis A, Psarros C, Triantafyllou C, Bendall J, Casadei B, Stefanadis C, Channon KM. Rapid, direct effects of statin treatment on arterial redox state and nitric oxide bioavailability in human atherosclerosis via tetrahydrobiopterin-mediated endothelial nitric oxide synthase coupling. Circulation. 2011 Jul 19;124(3):335-45. doi: 10.1161/CIRCULATIONAHA.110.985150. Epub 2011 Jul 5. PMID 21730307
- [Derived] Antoniades C, Bakogiannis C, Tousoulis D, Reilly S, Zhang MH, Paschalis A, Antonopoulos AS, Demosthenous M, Miliou A, Psarros C, Marinou K, Sfyras N, Economopoulos G, Casadei B, Channon KM, Stefanadis C. Preoperative atorvastatin treatment in CABG patients rapidly improves vein graft redox state by inhibition of Rac1 and NADPH-oxidase activity. Circulation. 2010 Sep 14;122(11 Suppl):S66-73. doi: 10.1161/CIRCULATIONAHA.109.927376. PMID 20837928